CLINICAL TRIAL: NCT07056608
Title: Comparison of Cardiovascular Disease Awareness in Patients With Rheumatoid Arthritis and Knee Osteoarthritis: A Cross-Sectional Study
Brief Title: Cardiovascular Disease Awareness in Rheumatoid Arthritis and Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 5.20.2025/approval no:4866
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Disease Risk; Rheumatoid Arthritis (RA); Knee Osteoarthritis
Keywords: Cardiovascular disease risk; rheumatoid arthritis; knee osteoarthritis; Cardiovascular Disease Risk Factors Knowledge Level
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis: Female patients aged 40 years and over with rheumatoid arthritis
- Knee osteoarthritis: Female patients aged 40 years and over diagnosed with knee osteoarthritis

SUMMARY:
Cardiovascular diseases (CVD) are still the most common cause of death. For these reasons, individuals, especially those with chronic diseases, need to be aware of CVD. CVD is also a significant cause of morbidity and mortality in rheumatoid arthritis (RA). This study aimed to compare CVD awareness in RA and knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
Patients who apply to our Physical Medicine and Rehabilitation clinic and are followed up with the diagnosis of RA and (KOA) will be screened. Demographic values such as age, gender, height, weight, smoking and alcohol use, diseases and medications used, cardiovascular disease awareness will be assessed with the Cardiovascular Disease Risk Factors Knowledge Level (CARRF-KL), exercise levels with the International Physical Activity Questionnaire (IPAQ), and nutritional habits with the Nutrition Attitude Scale (NAS). Cardiovascular risk calculation will be made with the Framingham Risk Score. It will also be ensured that patients with high risk are directed to the relevant branches. In addition, the Timed Up and Go Test (TUG), which is a prognosis indicator for cardiovascular diseases, will be performed. All surveys will be filled out in both groups and compared in terms of cardiovascular risk awareness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 and over
* Patients diagnosed with rheumatoid arthritis or osteoarthritis
* Volunteering to participate in the study

Exclusion Criteria:

* Patients who cannot ambulate
* Patients who cannot be evaluated due to cognitive reasons
* Those who are not receiving enteral nutrition or whose general condition is so poor that they cannot exercise

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with rheumatoid arthritis or knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Risk Factors Knowledge Level | Day 1
  This scale consists of 28 items. The first four items question the characteristics, protection and age factor of CVDs, 15 items question risk factors, and 9 items question the results of changes in risk behaviors. The items are answered as "Yes", "No" or "I don't know" and 1 point is given for each correct answer. The highest total score is 28. As the scores increase, the level of knowledge increases.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Day 1
  The short form of the questionnaire was used in this study. This short form consists of seven questions and provides information about the time spent in sitting, walking, moderate activities and vigorous activities. In activity assessment, the criterion is that each activity is performed for at least 10 minutes at a time. A score is obtained as "MET-min/week" by multiplying the time in minutes, the number of days and the MET value corresponding to the basal metabolic rate (multiples of resting oxygen consumption). Accordingly, the physical activity levels of the participants are classified as inactive, minimally active and very active according to the total physical activity score.
Nutrition Attitude Scale | Day 1
  The lowest score from the nutrition attitude scale is 21 and the highest score is 105. High scores from the scale indicate that individuals who fill out the scale have a high attitude towards nutrition, while individuals who receive low scores indicate that their attitude towards nutrition is low. It can be said that individuals with high attitude scores towards nutrition are sensitive to weight control and health.
Timed Up and Go Test | Day 1
  This test involves the individual getting up from a chair, walking 3 meters, returning and sitting on the chair. A stopwatch is kept during this process. If this time is 12 seconds or more, the individual is at risk of falling. This test is also used in cardiovascular disease risk assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Medical Doctor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital, İstanbul, Turkey
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided